CLINICAL TRIAL: NCT06293898
Title: A Phase 1 Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BL-M07D1 in Subjects With HER2 Expressing Advanced Malignant Solid Tumors
Brief Title: Open Label Study to Evaluate BL-M07D1 in HER2 Expressing Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-ST-101
Record Dates: First submitted 2024-02-22; First posted 2024-03-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; Cervical Cancer; Ovarian Cancer; Urothelial Carcinoma; Biliary Tract Cancer; Breast Cancer; Lung Cancer; Gastric Cancer; Gastroesophageal-junction Cancer; Esophageal Cancer
Keywords: HER2
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Carcinoma, Transitional Cell; Biliary Tract Neoplasms; Breast Neoplasms; Lung Neoplasms; Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: Dose Escalation (Experimental): Beginning with Cycle 1, BL-M07D1 will be administered on Day 1 by (IV) infusion every 3 weeks (D1Q3W)
  Interventions: Drug: BL-M07D1
- Experimental: Dose Finding (Experimental): Beginning with Cycle 1, BL-M07D1 will be administered on Day 1 by (IV) infusion every 3 weeks (D1Q3W)
  Interventions: Drug: BL-M07D1
- Experimental: Dose Expansion (Experimental): Beginning with Cycle 1, BL-M07D1 will be administered on Day 1 by (IV) infusion every 3 weeks (D1Q3W)
  Interventions: Drug: BL-M07D1

INTERVENTIONS:
Drug: BL-M07D1 — Drug: BL-M07D1 The study includes 3 parts: Part 1 Dose escalation. Part 2 Dose Finding non-randomized and Part 3 Dose expansion randomized. BL-M17D1 will be administered on Day 1 by intravenous infusion every 3 weeks.
  Other Names:
  BL-M07D1

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, and efficacy of BL-M07D1 in patients with HER2 expressing advanced tumors.

DETAILED DESCRIPTION:
BL-M07D1-ST-101 is a global, multi-center, Phase 1 study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of BL-M07D1 in participants with HER2 expressing advanced malignant solid tumors.

This study will be conducted in three parts (dose escalation, dose finding and dose expansion). Dosing will be conducted on Day 1 of a continuous 21-day treatment cycle. .

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years
2. Has a life expectancy of ≥3 months
3. Has documented locally advanced or metastatic HER2expressing (IHC 1+ to 3+ and/or HER2 gene amplification or activating mutation in tumor specimen by ISH or NGS) solid tumor(s) not amenable to curative surgery or radiation and has received at least 2 lines of standard therapy, including adjuvant/neoadjuvant treatment, or whose cancer is considered refractory to the standard of care or for which no standard treatment is available, including:

   1. Cohort 1: Subjects with HER2 expression in endometrial cancers (EC)
   2. Cohort 2: Subjects with HER2 expression in cervical cancers (CC)
   3. Cohort 3: Subjects with HER2 expression in ovarian cancers (OC) including fallopian tube cancer and primary peritoneal cancer
   4. Cohort 4: Subjects with HER2 expression in urothelial cancers (UC)
   5. Cohort 5: Subjects with HER2 expression in biliary tract cancers (BTC)
   6. Cohort 6: Subjects with HER2 expression in breast cancer (BC)
   7. Cohort 7: Subjects with HER2 expression in lung cancer (LC)
   8. Cohort 8: Subjects with HER2 expression in gastric, esophageal, or gastroesophageal junction (GEJ) cancers
4. Agree to provide most recent existing tumor samples (FFPE tissue block or slides) from primary or metastatic sites for tissue-based IHC staining to centrally determine HER2 expression:

   1. In dose escalation and dose finding: archival tissue or fresh biopsy. If no archival tissue is available, or it is not possible to obtain a fresh tissue biopsy, medical monitor approval is required to screen subject;
   2. In dose expansion: an FFPE block or slides from fresh biopsy or the most recent archival tissue is required.
5. Has at least one measurable lesion based on RECIST (Response Evaluation Criteria in Solid Tumors) V1.1
6. Has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1
7. Toxicity of previous antitumor therapy has returned to Grade ≤1
8. Has no serious cardiac dysfunction, left ventricular ejection fraction ≥50%
9. Has adequate organ function before enrollment, defined as:
10. Coagulation function: international normalized ratio (INR) ≤1.5×ULN, and activated partial thromboplastin time (APTT) ≤1.5 ULN, unless receiving anticoagulation therapy with prothrombin time and aPTT levels within the intended therapeutic range
11. Urinary protein ≤2+ or ≤1000 mg/24 hours
12. For premenopausal women with childbearing potential, a pregnancy test must be taken within 7 days prior to the start of treatment. Serum or urine pregnancy test must be negative and subject must be nonlactating.
13. Must agree to use adequate contraceptive measures during the treatment and for 6 months after the end of treatment for all subjects (regardless of gender)

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy, radical radiotherapy, targeted therapy (including small molecule inhibitor of tyrosine kinase), and other antitumor therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first administration; major surgery within 4 weeks prior to the first administration; mitomycin and nitrosoureas treatment within 6 weeks prior to the first administration
2. Subjects with history of severe heart disease
3. Subjects with prolonged QT interval (QTc >470 msec), complete left bundle branch block, Grade 3 atrioventricular block
4. Active autoimmune diseases and inflammatory diseases
5. Other malignant tumors diagnosed within 3 years prior to the first administration considered to be in remission
6. Subjects with poorly controlled hypertension by 2 types of antihypertensive drugs (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg)
7. Subjects with advanced or clinically significant lung diseases, such as poorly controlled chronic obstructive pulmonary disease and asthma, restrictive lung disease, pulmonary hypertension, etc.
8. Subjects with stroke, transient ischemic attack within 6 months before enrollment
9. Subjects with a thromboembolic event (eg, deep vein thrombosis [DVT] or pulmonary embolism [PE]) within 6 months before enrollment except for those who are clinically stable and receiving treatment with adequate anticoagulant therapy for at least 3 weeks before enrollment
10. Patients with primary tumors in the central nervous system (CNS) and active or untreated CNS metastases and/or carcinomatous meningitis should be excluded. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks and have no evidence of new or enlarging brain metastases and no requirements for corticosteroids 14 days prior to dosing with the investigational product (IP). Patients on low dose corticosteroids (<20 mg prednisone or equivalent/day) may participate.
11. Subjects with pre-existing Grade ≥2 peripheral neuropathy Subjects who have a history of allergies to recombinant humanized antibodies or human-mouse chimeric antibodies or any of the components of BL M07D1

11. Subjects who are receiving treatment with systemic glucocorticoids >10 mg/day equivalent of prednisone, except for the treatment of chronic obstructive pulmonary disease, antiemetic, infusion reactions; however, treatment with low dose glucocorticoids (≤10 mg/day equivalent of prednisone) is permitted. The chronic use of topical, inhaled, and locally injected steroids is permitted 12. Subjects who have received treatment with anthracyclines with a cumulative dose exceeding 360 mg/m2 13.Subjects with known human immunodeficiency virus (HIV) infection (HIV antibody positive). Subjects are allowed to participate if all the following criteria are met:

1. Undetectable HIV RNA and CD4 count ≥ 350 cells/μL at screening;
2. No AIDS-defining opportunistic infection within 12 months prior to screening;
3. On stable antiretroviral therapy (ART) for at least 4 weeks prior to enrollment with projected continuation of ART as clinically indicated while on the study.

   14. Subjects with known active hepatitis C virus (HCV) infection (HCV antibody positive and HCV-RNA > the lower limit of detection). Subjects with a positive anti-HCV antibody are eligible only if PCR is negative for HCV RNA 15. Subjects with known active tuberculosis 16 .Subjects with active infections requiring IV antibiotic, antiviral, or antifungal treatment, such as severe pneumonia, bacteremia, sepsis, etc., within 1 week prior to first dose of study treatment. Subjects on stable oral antimicrobials with no clinical or laboratory evidence of active infection are eligible.

   17. Subjects who are pregnant or, breastfeeding, or planning to become pregnant during the study 18. Other conditions that the investigator or sponsor believes are not suitable for participating in this clinical trial.

   16. Other conditions that the investigator believes are not suitable for participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Summary of safety | Though study completion, an average of 24 months
  The number of patients with dose-limiting toxicities, serious adverse events, treatment-emergent adverse events, physical exam findings, vital signs, laboratory tests, ECG parameters and echocardiograph
To determine the maximum tolerated dose (MTD) if reached or maximum administered dose (MAD) and two or more recommended doses for dose expansion (RDEs) of BL-M07D1 | 21 Days
  Determine the highest BL-M07D1 dose level at which subjects do not experience a DLT during the DLT evaluation period and highest BL-M07D1 dose administered in the event and MTD cannot be defined.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Leader, Study Director — SystImmune Inc.
Locations (17):
- United States (17):
  - University of Alabama Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Cedars Sinai, Los Angeles, California
  - Scripps Health, San Diego, California
  - University of Miami, Miami, Florida
  - Sarah Cannon Research institute - Lake Nona Florida, Orlando, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institiute, Detroit, Michigan
  - NYU Langone Hospital - Long Island Investigational Pharmacy, Mineola, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Oncology Consultants, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia